CLINICAL TRIAL: NCT03711188
Title: A Study of the Safety and Efficacy of IMM-101 in Combination With Checkpoint Inhibitor Therapy in Patients With Advanced Melanoma
Brief Title: A Study of IMM-101 in Combination With Checkpoint Inhibitor Therapy in Advanced Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Immodulon Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMM-101-015
Record Dates: First submitted 2018-10-04; First posted 2018-10-18 (Actual); Results first posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2023-11

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Ipilimumab; IMM-101

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMM-101 (and nivolumab or ipilimumab) (Experimental): Patients in cohort A were given IMM-101 in combination with nivolumab. Patients in cohort B who fail to respond to treatment with IMM-101 and nivolumab, and who meet certain criteria, have the option to change treatment on study to IMM-101 and ipilimumab.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: IMM-101

INTERVENTIONS:
Drug: Nivolumab — Nivolumab is to be administered as a 3 mg/kg IV infusion every two weeks in accordance with the prescribing information.
  Other Names: Opdivo
Drug: Ipilimumab — Ipilimumab, when used as subsequent treatment for patients in cohort B, is to be administered as a 3 mg/kg IV infusion over 90 minutes every three weeks for a maximum of 4 doses, in accordance with the prescribing information.
  Other Names: Yervoy
Drug: IMM-101 — A single 0.1 mL intradermal injection of IMM 101 (10 mg/mL) given every 2 weeks for the first 3 doses followed by a rest period of 4 weeks, then one dose every 2 weeks for the next 3 doses. This is followed by a dose every 4 weeks thereafter.
  Other Names: Heat killed whole cell M. obuense National Collection of Type Cultures (NCTC) 13365

SUMMARY:
The purpose of this study is to assess the safety and efficacy of the combination of IMM-101 with nivolumab.

DETAILED DESCRIPTION:
This open-label study will assess the safety and efficacy of the combination of IMM-101 with nivolumab in patients with unresectable stage III, or stage IV melanoma who are either treatment-naive (cohort A) or whose disease has progressed during PD-1 blockade (cohort B). Ipilimumab may be used as a subsequent treatment in place of nivolumab alongside IMM-101 for patients in cohort B if their disease progresses on study. Eighteen patients will be enrolled into cohort A and 8 patients into cohort B.

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically-confirmed diagnosis of advanced (unresectable Stage III) or metastatic (Stage IV) melanoma.
2. At least one measurable lesion by CT or MRI, according to RECIST 1.1.
3. Eastern Cooperative Oncology Group (ECOG)/World Health Organisation (WHO) Performance Status of ≤1 at Day 0.
4. Known BRAF V600 mutation status or consent to BRAF V600 mutation testing during the Screening Period.
5. Prior radiotherapy must have been completed at least 2 weeks prior to study drug administration (Week 0, Visit 1). Prior adjuvant or neoadjuvant melanoma therapy is permitted if it was completed at least 6 weeks prior to enrolment (Week 0, Visit 1), and all related adverse events have resolved or stabilised.
6. Patient is considered suitable for treatment with nivolumab.

For cohort A, the following key inclusion criteria apply:

1. Patient is treatment-naive (i.e. no prior systemic anticancer therapy for unresectable or metastatic melanoma).

For cohort B, the following key inclusion criteria apply:

1. Patient is either currently receiving treatment with an anti-PD-1 therapy (monotherapy or in combination with ipilimumab), for advanced melanoma and has progressive disease by RECIST 1.1 after 4 or more doses; or has previously received at least 4 doses of PD-1 targeted therapy, alone or in combination with ipilimumab, had disease progression by RECIST 1.1 during this therapy and has not received any further therapy for advanced melanoma.

Key Exclusion Criteria:

1. Uveal/ocular melanoma.
2. Active brain metastases or leptomeningeal metastases. Patients with brain metastases are eligible for cohort B of the study only, if these have been treated and there is no MRI evidence of progression for at least 8 weeks after treatment is complete and within 21 days prior to first dose of study treatment administration.
3. Patient has documented history of clinically severe autoimmune disease or a syndrome that requires systemic steroids or immunosuppressive agents.
4. Patient has a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or immunosuppressant drugs (such as azathioprine, tacrolimus, cyclosporin) within the 14 days period before the first administration of IMM-101.

For cohort A, patients meeting the following key criteria are also ineligible to participate in this study:

1. Patient has received prior therapy with an anti-programmed cell death-1 (anti-PD-1), anti-PD ligand-1 (PD-L1), anti-PD-L2, anti-CD137 antibody, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) agent.

For cohort B, patients meeting the following key criteria are also ineligible to participate in this study:

1. Patient has received more than one treatment regimen for advanced (stage III/IV) disease prior to their anti PD-1 therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Fusi, Principal Investigator — St George's University Hospitals NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - St George's University Hospitals NHS Foundation Trust, London
  - The Christie Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty-two patients at 2 centres were consented and screened. Six patients failed to meet one or more of the specific inclusion criteria or met one or more exclusion criteria and were deemed screen failures.
Period: Overall Study
Arm/Group | IMM-101 (and Nivolumab or Ipilimumab)
Started | 16
Completed | 4
Not Completed | 12
Not completed — Disease progression | 11
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all patients with confirmation of eligibility at Screening.
Arm/Group | IMM-101 (and Nivolumab or Ipilimumab)
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 10
Age, Continuous [Median (Full Range); unit: years] | 68.5 [36 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 16
PD-L1 status in Cohort A patients only [Number; unit: participants] — Subgroups of patients in cohort A (n=11) were defined based on PD-L1 status (PD-L1 positive and PD-L1 negative/indeterminate) at Screening. For one patient PD-L1 status was unknown. Population: PDL-1 status was only determined in Cohort A patients (n=11) thus the Row population differs from the Overall population (n=16).
  participants
    PD-L1 Positive: number analyzed (Participants) | 11
    PD-L1 Positive | 6
    PD-L1 Negative or Indeterminate: number analyzed (Participants) | 11
    PD-L1 Negative or Indeterminate | 4
    PD_L1 status Not Assessed or Unknown: number analyzed (Participants) | 11
    PD_L1 status Not Assessed or Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of the Combination of IMM-101 + Nivolumab
Description: Incidence, frequency and severity of treatment emergent adverse events (TEAEs) throughout the study.
Time Frame: From the point of Informed Consent until end of the study assessment (up to 84 weeks) or until withdrawal from the study.
Population: The Safety Analysis Set (SAF) included all patients who received at least one dose of IMM-101, irrespective of compliance with eligibility and other protocol criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | IMM-101 (and Nivolumab or Ipilimumab)
Number analyzed (Participants) | 16
Participants
  Treatment emergent adverse events (TEAEs) | 16
  Treatment-related TEAEs | 14
  Serious TEAEs | 6
  Immune relared TEAEs | 14
  TEAEs leading to discontinuation of IMM-101 | 3
  TEAEs leading to withdrawal | 1
  TEAEs leading to death | 0

2. Primary Outcome: Overall Response Rate
Description: The primary endpoint of Overall Response Rate (ORR) is defined as the number of subjects with a Best Overall Response (BOR) of confirmed Complete Response (CR) or Partial Response (PR) divided by the number of subjects in the Intent-to-treat analysis set in each cohort of the study.
  The BOR will be determined once all the data up to and including the 12-month assessments for Cohort A or the 6-month assessment for Cohort B are available. It is defined as the best response designation based on confirmed responses determined by the investigator according to RECIST 1.1, recorded between the date of first postscreening scan and the date of last scan at/prior to the assessment at the 12-month assessment (Cohort A) and 6-month assessment/last assessment prior to change of treatment to IMM-101 + ipilimumab whichever is sooner (Cohort B).
Time Frame: From enrollment to end of study (18 months) or withdrawal, whichever was soonest
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A: Patients in cohort A were treatment-naive and were required to have had a tumour sample (archived tissue in the last 3 months or newly obtained biopsy) that was adequate for PD-L1 assessment prior to enrolment.
  These 11 patients received IMM-101 in addition to Nivolumab.
- Cohort B: Patients in cohort B were either currently on (or had previously received) treatment with an anti-PD-1 therapy (monotherapy or in combination) for advanced melanoma and had progressive disease by RECIST 1.1 after at least 3 doses of anti-PD-1 given as monotherapy or at least 2 doses of anti-PD-1 given in combination regimes and had not received any therapy since for advanced melanoma.
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 5
Participants | 8 | 0

3. Secondary Outcome: Best Overall Response (BOR) Using RECIST 1.1
Description: Best Overall Response (BOR) is defined as the best response (complete or partial response, stable disease or progressive disease) designation based on confirmed responses determined by the investigator according to RECIST 1.1, recorded between the date of first postscreening scan and the date of last scan at/prior to the assessment at the 12-month assessment (Cohort A) and 6-month assessment/last assessment prior to change of treatment to IMM-101 + ipilimumab whichever is sooner (Cohort B).) Patients in cohort B who changed therapy without documented progression were censored at their last scan assessment prior to the change of therapy.
Time Frame: 18 months
Population: Intent to treat population - all patients who received at least one dose of IMM-101
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 5
Participants
  Complete Response (CR) | 2 | 0
  Partial Response (PR) | 6 | 0
  Stable Disease | 1 | 0
  Disease Progression | 2 | 5

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival was defined as the time from Visit 1 (week 0) to the first confirmation of progression using RECIST 1.1 (confirmed or unconfirmed), or death from any cause (whichever occurred first). Progression was determined by the investigator using the CT or MRI scan or death due to any cause. Patients who died without reporting progression were considered to have progressed on the date of their death. Progression is defined by RECIST 1.1 guidelines as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: From Visit 1 (week 0) and the first confirmation of progression using RECIST 1.1 (confirmed or unconfirmed), or death from any cause (whichever occurred first).
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 5
Participants
  Less than or equal to 3 months | 2 | 4
  >3 months but < or = to 6 months | 1 | 1
  >6 months but < or = to 9 months | 3 | 0
  >9 months but < or = to 12 months | 1 | 0
  >12 months but < or = to 18 months | 0 | 0
  .18 months | 4 | 0

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from Visit 1 (week 0) until date of death from any cause. OS was calculated for the entire study duration, where patients without a death date were right censored at the date the patient was last known to be alive. Post-study survival information was collected until database lock, for subjects completing or withdrawing from the study and included in the analysis.
Time Frame: Overall survival was defined as the time from Visit 1 (week 0) until the end of the study (80 weeks) or until the date of death from any cause.
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 5
Participants
  < or = to 3 months | 1 | 0
  >3 months but < or = to 6 months | 0 | 0
  >6 months but < or = to 9 months | 1 | 2
  >9 months but < or = to 12 months | 0 | 2
  >12 months but < or = to 18 months | 0 | 1
  >18 months | 9 | 0

6. Secondary Outcome: Overall Survival (OS) at One Year
Description: Number of patients surviving at leat 12 months
Time Frame: OS at 1 year was calculated after all patients had had the opportunity of 12 months treatment of study
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 5
Participants | 9 | 1

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) were recorded on the patient's electronic case report form (eCRF) from the time of informed consent until the end of study (18 months later) . All AEs were followed until resolution, death, or 30 days after the last administration of study treatment (whichever came first).
Description: Incidence, frequency and severity of treatment-emergent adverse events (TEAEs; all TEAEs, serious adverse events (SAEs), treatment-related TEAEs, immune-related AEs, and TEAEs leading to IMM-101 discontinuation or study withdrawal).
Groups:
- IMM-101 and Nivolumab: * Patients in Cohort A were initially treated with IMM-101 and nivolumab.
  * Patients in Cohort B were initially treated with IMM-101 + nivolumab and when they failed to respond to nivolumab they had the option to switch treatment.
  Nivolumab was administered as a 3 mg/kg IV infusion every two weeks in accordance with the prescribing information.
- IMM-101 and Ipilimumab: • Patients from Cohort B who failed to respond to nivolumab and met certain criteria had the option to switch to ipilimumab.
  Ipilimumab, when used as subsequent treatment for patients in Cohort B, was administered as a 3 mg/kg IV infusion over 90 minutes every three weeks for a maximum of 4 doses, in accordance with the prescribing information.
Arm/Group | IMM-101 and Nivolumab | IMM-101 and Ipilimumab
All-Cause Mortality (participants affected / at risk) | 8/16 | 1/1
Serious Adverse Events (participants affected / at risk) | 12/16 | 1/1
Other Adverse Events (participants affected / at risk) | 16/16 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMM-101 and Nivolumab (N=16) | IMM-101 and Ipilimumab (N=1)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Epistaxis (Blood and lymphatic system disorders) | 1 (1) | 0
Pyrexia (General disorders) | 1 (1) | 0
Chills (General disorders) | 1 (1) | 0
Fatigue (General disorders) | 1 (1) | 0
Lethargy (General disorders) | 1 (1) | 0
Pain (General disorders) | 1 (1) | 0
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Wrist fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Spinal cord compression (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Cortisol deficiency (Endocrine disorders) | 1 (1) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMM-101 and Nivolumab (N=16) | IMM-101 and Ipilimumab (N=1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 7 (9) | 0 (0)
Fatigue (General disorders) | 6 (9) | 0 (0)
Injection site erythema (General disorders) | 4 (6) | 0
Pruritis (General disorders) | 4 (5) | 0 (0)
Injection site swelling (General disorders) | 3 (5) | 0 (0)
Injection site ulcer (General disorders) | 3 (4) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
influenza like illness (General disorders) | 1 (1) | 0 (0)
Injection site vesicles (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Bartholins cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Nervous system disorders) | 2 (3) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (4) | 1 (1)
Breath odour (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth Ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 4 (4) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Coronavirus test positive (Investigations) | 1 (1) | 0 (0)
Haemoglobin deecresed (Investigations) | 1 (1) | 0 (0)
Vitamin D decreased (Investigations) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Oral infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The Overall Response Rate shows encouraging results in Cohort A with 73% of responses confirmed by subsequent scans (18% patients had a BOR (RECIST 1.1) of complete response (CR) and 55% of partial response (PR)). Limitations are the small sample size. This finding would need to be confirmed in a larger trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/88/NCT03711188/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/88/NCT03711188/SAP_001.pdf